CLINICAL TRIAL: NCT00307944
Title: Randomized, Placebo-Controlled Trial of Pantoprazole for Sleepiness Associated With Acid Reflux and Obstructive Sleep Disordered Breathing
Brief Title: Study of Pantoprazole for Sleepiness Associated With Acid Reflux and Sleep Apnea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 04-06-24-04
Record Dates: First submitted 2006-03-27; First posted 2006-03-28 (Estimated); Last update posted 2007-12-12 (Estimated); Status verified 2007-12

CONDITIONS: Acid Reflux Disease; Obstructive Sleep Apnea
Keywords: Acid Reflux; Obstructive Sleep Apnea; Daytime Sleepiness
MeSH Terms: conditions — Gastroesophageal Reflux; Sleep Apnea, Obstructive; Disorders of Excessive Somnolence | interventions — Pantoprazole

INTERVENTIONS:
Drug: Pantoprazole

SUMMARY:
The purpose of this study is to determine if using Pantoprazole decreases your daytime sleepiness and improves your reaction time when compared to using a placebo (sugar pill).

DETAILED DESCRIPTION:
Half of the patients enrolled in the study will begin the study taking Pantoprazole. The other half will begin the study taking a placebo (sugar pill). There is an equal chance of being placed in either group.

After two weeks, the patients will stop taking their first batch of medication to allow it to completely leave their bodies. Then the patients will begin taking the other medication so that by the end of the study, each patient will have been treated with pantoprazole for two weeks and placebo for two weeks.

At the end of each two weeks, patients will be asked to complete questionnaires regarding their daytime sleepiness and reflux symptoms. Patients will also complete reaction time testing as a measure of daytime sleepiness.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Daytime sleepiness (ESS >= 8)
* Mild to moderate OSD (AHI<=30)
* Symptoms of GERD
* Symptoms of acid reflux

Exclusion Criteria:

* Pregnant or trying to become pregnant
* Depression or unstable psychiatric disorder
* Allergy to Pantoprazole
* Taking a proton pump inhibitor within the last month
* Taking a histamine-2 receptor blocker within the last month
* Automobile or industrial accident due to daytime sleepiness
* Currently taking ketoconazole, itraconazole, ampicillin or iron salts
* Hypersecretory acid disorder (Zollinger-Ellison Syndrome)
* Active peptic ulcer disease
* Severe concomitant disease of another major body system
* Malignancy in the past 5 years
* Current abuse of alcohol, medication or drugs
* Sedative medications
* Additional treatment for obstructive sleep apnea (i.e. CPAP or surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68
Dates: Start 2004-08; Study Completion 2006-08

PRIMARY OUTCOMES:
Difference between treatment groups with regard to change in sleepiness score (ESS)

SECONDARY OUTCOMES:
Difference between treatment groups with regard to change in reaction time testing.
Difference between treatment groups with regard to change in total reflux symptom scores.
Difference between treatment groups with regard to change in sleep related QOL (FOSQ).

CONTACTS AND LOCATIONS:
Overall Officials: David L Steward, MD, Principal Investigator — University Ear, Nose and Throat Specialists
Locations (1):
- University Ear, Nose and Throat Specialists, Cincinnati, Ohio, United States